CLINICAL TRIAL: NCT04636073
Title: A Prospective, Multicenter, Non-randomized, Single-arm, Open-label Clinical Study to Demonstrate the Safety and Performance of the Leaflex™ Performer
Brief Title: The Leaflex™ Early Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Reprioritization of attention and resources by Sponsor.
Sponsor: Pi-cardia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02-CLN-028
Record Dates: First submitted 2020-10-30; First posted 2020-11-19 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2024-05

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Leaflex™ Performer (Experimental)
  Interventions: Device: Leaflex™ Performer

INTERVENTIONS:
Device: Leaflex™ Performer — A transfemoral catheter designed to treat calcific aortic stenosis by scoring the calcification in the aortic valve leaflets.

SUMMARY:
A prospective, multicenter, single-arm, early feasibility study aimed to assess safety and performance of the Leaflex™ Performer in the treatment of patients with symptomatic, severe aortic stenosis.

DETAILED DESCRIPTION:
A prospective, multicenter, single-arm, early feasibility study aimed to assess safety and performance of the Leaflex™ Performer in the treatment of patients with symptomatic, severe aortic stenosis.

Subjects will be seen at pre- and post procedure, discharge, 30 days and at 3, 6, 9 and 12 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptomatic, severe aortic stenosis who are operable, but not recommended by the heart team for immediate treatment with surgical or transcatheter aortic valve replacement.
* Patient is willing to comply with scheduled visits and tests and is able and willing to provide informed consent.

Exclusion Criteria:

* Inoperable for emergency surgery.
* Moderate or greater aortic regurgitation.
* Anatomic contraindications.
* Coronary, carotid, or vertebral artery disease that, in the opinion of the heart team, should be treated; or treatment of coronary artery disease ≤ 1 month prior to index procedure.
* Aortic balloon valvuloplasty ≤ 3 months prior to index procedure.
* Stroke ≤ 12 months prior to index procedure.
* History of a myocardial infarction ≤ 6 weeks prior to index procedure.
* Patients with clinically significant abnormality in cell blood count, history of bleeding diathesis or coagulopathy.
* Hemodynamic instability.
* Hypertrophic cardiomyopathy with obstruction.
* Left ventricle ejection fraction <30%.
* Ongoing severe infection, including endocarditis, or sepsis.
* Life expectancy ≤ 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in aortic valve area | Baseline to 3 days
  assessed by echo

SECONDARY OUTCOMES:
Rate of all-cause mortality and all-cause stroke (VARC 2) | 30 days post procedure
  Composite
Rate of worsening of aortic regurgitation | Baseline to 30 days
  by greater than 1 grade
Rate of worsening of aortic regurgitation | Discharge to 30 days
  by greater than 1 grade
Rate of device related adverse events | 12 months
Change in 6 minute walk test | 1, 6 and 12 months
  distance (meters)
Quality of Life Improvement | 1, 6 and 12 months
  measured by KCCQ
Quality of Life Improvement | 1, 6 and 12 months
  measured by EQ5D
Change in aortic valve area | 30 day, 3, 6, 9, 12 months
  assessed by echo
Change in pressure gradients | 30 day, 3, 6, 9, 12 months
  assessed by echo